CLINICAL TRIAL: NCT00751686
Title: To Estimate the Burden of Rotavirus Gastroenteritis (RV GE) in Children < 5 Years of Age in Greece
Brief Title: Estimation of the Burden of Rotavirus Gastroenteritis (RV GE) in Children Less Than 5 Years in Greece
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 109355
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Rotavirus Gastroenteritis
Keywords: Gastroenteritis; Burden; Rotavirus; < 5 years; Greece; Children
MeSH Terms: conditions — Gastroenteritis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample

GROUPS / COHORTS (1):
- RV GE Group
  Interventions: Procedure: Stool sample; Other: Data collection

INTERVENTIONS:
Procedure: Stool sample — Collection of the stool at least 48 hours after hospitalisation. Stool samples should be obtained preferably within 4 and no later than 10 days after the onset of the GE symptoms.
Other: Data collection — Logbook, Health Economic Questionnaire, Telephone call.

SUMMARY:
The purpose of this study is to measure the disease burden from RV GE among children less than 5 years of age using hospital surveillance data. In addition, data collected will determine the seasonal distribution, disease severity, age distribution of RV GE. From an economic standpoint, the cost and impact of RV will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child < 5 years of age at the time of the visit (a child becomes ineligible on the day of her/his 5th birthday).
* Child is brought to the emergency room for acute GE during the study period or develop acute GE at least 48 hours after hospitalisation.
* Written informed consent obtained from the parent/guardian of the subject.
* Children with RV positive stool sample will be enrolled in the study.

Exclusion Criteria:

• Not applicable.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children < 5 years of age seen at the selected hospital sites for acute GE (e.g. subjects treated at the hospital or visiting the emergency room for an acute GE episode or developed acute GE at least 48 hours after hospitalisation) with a rapid screen positive test result to RV.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Estimation of the proportion of RV GE among all acute GE emergency room visits among children <5 years of age. | Approximately 12 months
Estimation of the proportion of RV GE among all acute GE hospitalisations among children <5 years of age. | Approximately 12 months
Estimation of the incidence of nosocomial RV GE among all hospitalised children <5 years of age. | Approximately 12 months

SECONDARY OUTCOMES:
Determination of the age of the children, disease severity, and the seasonal distribution of RV GE among children <5 years of age. | Approximately 12 months
Assessing the costs related to the episodes of RV GE, by the completion of the Health Economic Questionnaire (interview with the parent for a subset of subjects) and the cost checklist provided by the hospital's site staff. | Approximately 12 months
Identification of prevalent genotypes of RV among children <5 years of age. | Approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Rio/Patras
  - GSK Investigational Site, Thessaloniki

REFERENCES:
- [Derived] Konstantopoulos A, Tragiannidis A, Fouzas S, Kavaliotis I, Tsiatsou O, Michailidou E, Spanaki A, Mantagos S, Kafetzis D, Papaevangelou V, Gopala K, Holl K. Burden of rotavirus gastroenteritis in children <5 years of age in Greece: hospital-based prospective surveillance (2008-2010). BMJ Open. 2013 Dec 11;3(12):e003570. doi: 10.1136/bmjopen-2013-003570. PMID 24334153